CLINICAL TRIAL: NCT00794898
Title: Onset of Efficacy of Anti-TNF Chimeric Monoclonal Antibody (Remicade) in the Treatment of Patients With Active Rheumatoid Arthritis Despite Methotrexate Treatment
Brief Title: Efficacy of Remicade in the Treatment of Active Rheumatoid Arthritis Despite Methotrexate (Study P03027)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03027
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Remicade in the treatment of patients with active RA despite treatment with MTX.
  Interventions: Biological: Infliximab (Remicade)

INTERVENTIONS:
Biological: Infliximab (Remicade) — Infliximab 3 mg/kg infusions at Weeks 0, 2, and 6. All patients will continue to receive the same dose of MTX they were receiving at entry throughout the subsequent treatment period.
  Other Names: Remicade; SCH 215596

SUMMARY:
This is an open-label program of Remicade in the treatment of patients with active rheumatoid arthritis (RA) despite treatment with methotrexate (MTX) to determine the onset of efficacy of infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, >=18 to <=75 years of age.
* Diagnosis of RA according to the revised 1987 criteria of the American Rheumatism Association (Arnett et al., 1988). The disease should have been diagnosed at least 6 months prior to Screening.
* Patients have active disease, in the opinion of the physician, despite the concomitant use of DMARDS. Evidence of active disease may include any of the following:

  6 or more swollen or tender joints; and 2 of the following
  * Morning stiffness >45 minutes
  * C-reactive protein >2.0 mg/L
  * ESR >28 mm/h
* Patients must have been using oral or parenteral MTX for at least 2 months with no break(s) in treatment of more than 2 weeks total during this period. Patients must have been on a stable dose of >=7.5 mg/wk (IM, SQ, PO) for at least 8 weeks prior to Screening.
* Men and women of childbearing potential must be using adequate birth control measures (abstinence, oral contraceptives, IUD, barrier method with spermicide or, surgical sterilization) and should continue such precautions for 6 months after receiving the last infusion.
* Patients must be on a stable dose of folic acid prophylaxis for at least 4 weeks prior to Screening.
* Patients using oral corticosteroids or NSAIDs, must have been on a stable dose for at least 4 weeks prior to Screening, and must continue during the treatment period. If currently not using corticosteroids or NSAIDs, the patient must have not received corticosteroids or NASIDs for at least 4 weeks prior to Screening.
* Patients must be able to adhere to the program visit schedule and other protocol requirements.
* Patients must be capable of giving informed consent and the consent must have been obtained prior to any screening procedures.

Exclusion Criteria:

* Pregnant women, nursing mothers or a planned pregnancy within 1.5 years of enrollment
* Patients who are incapacitated, largely or wholly bedridden or confined to a wheelchair, and who have little or no ability for self-care.
* Patients who have any current systemic inflammatory condition with signs and symptoms that might confound the evaluations of benefit from the Remicade therapy, eg, Lyme disease, or a rheumatic disease other than RA.
* Use of DMARDS other than MTX within 4 weeks prior to Screening.
* Use of intra-articular, IM, or IV. corticosteroids (including IM ACTH) within 4 weeks prior to Screening.
* Prior administration any other therapeutic agent targeted at reducing TNF (eg, Etanercept, pentoxifylline, thalidomide or anti-CD4+ antibody) within the previous 6 months.
* Treatment with any investigational drug within the previous 6 months.
* A history of known allergies to murine proteins.
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months. Less serious infections in the previous 3 months, such as acute upper respiratory tract infection (colds) or uncomplicated urinary tract infection need not be considered exclusions at the discretion of the treating physician.
* History of opportunistic infections such as herpes zoster within 2 months of Screening. Evidence of active CMV, active pneumocystis carinii, drug resistant atypical mycobacterium, etc.
* Documented HIV infection.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
* Any currently known malignancy or pre-malignant lesions or any history of malignancy within the past 5 years.
* Patients with alcoholism, alcoholic liver disease, or other chronic liver disease.
* Patients with a positive PPD within 3 months and chest X-Ray suggestive of active TB or a previous exposure to TB.
* Patients with CHF, even if asymptomatic or not requiring medication must be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-07-01 (Actual); Primary Completion 2004-04-01 (Actual); Study Completion 2004-04-01 (Actual)

PRIMARY OUTCOMES:
Define the onset of efficacy of infliximab in patients with active RA, using the validated SF-36 questionnaire. | After the first 2 weeks of treatment.

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html